CLINICAL TRIAL: NCT06968585
Title: A Phase III,Multicenter,Randomized,Open-Label,Active-Controlled Trial of A166 Versus Trastuzumab Emtansine (T-DM1) in Patients With HER2-Positive Unresectable or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane Therapy
Brief Title: A Study of A166 Versus Trastuzumab Emtansine (T-DM1) in Patients With HER2-Positive Unresectable or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane Therapy
Acronym: A166
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KL166-III-06
Record Dates: First submitted 2025-04-26; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A166 (Experimental): A166 is administered intravenously at a dose of 4.8 mg/kg every 21 (±3) days (q3w).
  Interventions: Drug: A166
- T-DM1 (Active Comparator): T-DM1 is administered intravenously at a dose of 3.6 mg/kg every 21 (±3) days (q3w).
  Interventions: Drug: T-DM1

INTERVENTIONS:
Drug: A166 — intravenous(IV) infusion (Q3W)
  Arms: A166
Drug: T-DM1 — intravenous(IV) infusion (Q3W)
  Arms: T-DM1

SUMMARY:
Evaluation of the efficacy of A166 versus trastuzumab emtansine (T-DM1) in Patients with HER2-Positive unresectable or metastatic breast cancer previously treated with trastuzumab and taxane therapy

DETAILED DESCRIPTION:
This study will evaluate the efficacy of A166 versus trastuzumab emtansine (T-DM1) in patients with HER2-positive unresectable or metastatic breast cancer previously treated with trastuzumab and taxane therapy

To further evaluate the efficacy of A166 versus T-DM1 in patients with HER2-positive unresectable or metastatic breast cancer, based on effectiveness endpoints including:

Overall survival (OS)

Progression-free survival (PFS) as assessed by investigators

Objective response rate (ORR), disease control rate (DCR), duration of response (DOR), and clinical benefit rate (CBR) assessed by both blinded independent central review (BICR) and investigators.

To assess the safety profile of A166 for injection in patients with HER2-positive unresectable or metastatic breast cancer.

To evaluate the immunogenicity of A166 for injection in patients with HER2-positive unresectable or metastatic breast cancer.

To characterize the pharmacokinetic (PK) profile of A166 for injection in patients with HER2-positive unresectable or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥ 18 years and ≤ 75 years when signing the informed consent form.
2. Breast cancer patients by histopathology and/or cytology documented.
3. Disease progression after receiving a trastuzumab-based regimen (or a commercially available trastuzumab biosimilar or inetetamab) in the advanced or metastatic setting, or disease progression/recurrence within 12 months during or after (neo)adjuvant therapy (with a trastuzumab-based regimen or commercially available trastuzumab biosimilar).
4. Have previously received taxanes.
5. Patients must have experienced disease progression or intolerance during or after the most recent treatment prior to randomization.
6. At least one measurable lesion according to RECIST 1.1 criteria

Exclusion Criteria:

1. Previous treatment with A166 or any HER2-targeted antibody-drug conjugate (ADC) with a microtubule inhibitor payload.
2. Known history of severe hypersensitivity to other monoclonal antibodies, or allergy to A166 , T-DM1 (trastuzumab emtansine) or their components.
3. Permanent discontinuation of trastuzumab or its biosimilars due to any toxicity in prior treatments.
4. Presence of severe corneal epithelial disease at baseline; or inability to perform daily activities without contact lenses.
5. Presence of spinal cord compression or clinically active central nervous system (CNS) metastases.
6. Other conditions considered by the investigator to make the patient unsuitable for participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Randomization up to approximately 39 months
  PFS as assessed by BICR according to RECIST v 1.1

SECONDARY OUTCOMES:
Overall survival (OS) | Randomization up to approximately 48 months
  OS, 1-year survival rate, 2-year survival rate, and 3-year survival rate.
Objective response rate(ORR) | Randomization up to approximately 39 months
  ORR is defined as the percentage of patients who achieve complete response(CR) or partial response (PR), as assessed by BICR/investigator per RECIST 1.1
Disease control rate(DCR) | Randomization up to approximately 39 months
  DCR is defined as the percentage of patients who achieve CR, PR or stable disease (SD), as assessed by BICR/investigator per RECIST 1.1
Duration of response(DOR) | Randomization up to approximately 39 months
  DoR is defined as the time from the date of first documented CR or PR until date of documented disease progression per RECIST 1.1, as assessed by BICR/investigator or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No